CLINICAL TRIAL: NCT04797403
Title: Effectiveness of Implementing an Intensive Blood Pressure Reduction Intervention on Cognitive Decline in Low-Income and Minority Hypertensive Patients
Brief Title: Implementation of Multifaceted Patient-Centered Treatment Strategies for Intensive Blood Pressure Control in Minimize Cognitive Decline
Acronym: IMPACTS-MIND
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Collaborators: Wake Forest University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Katherine T Mills, Assistant Professor, Tulane University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R61AG068481 (NIH); R33AG068481 (NIH)
Record Dates: First submitted 2021-03-08; First posted 2021-03-15 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Hypertension; Cognitive Decline
MeSH Terms: conditions — Hypertension; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Cluster-randomized trial with randomization at the clinic level
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The core component of the intervention is protocol-based treatment using the SPRINT intensive BP management algorithm. Implementation strategies include dissemination of SPRINT study findings, team-based collaborative care and shared-decision making, blood pressure audit and feedback, home blood pressure monitoring, and health coaching.
  Interventions: Behavioral: Stepped-care protocol adapted from the SPRINT intensive-treatment algorithm
- Enhanced Usual Care (No Intervention): Enhanced usual care will include an education session on the ACC/AHA hypertension guideline to providers and proper BP measurement to providers and staff at enhanced usual care clinics.Otherwise, no active intervention will take place, and all usual care clinics will follow their routine clinic practice.

INTERVENTIONS:
Behavioral: Stepped-care protocol adapted from the SPRINT intensive-treatment algorithm — The core component of the intervention is protocol-based treatment using the SPRINT intensive BP management algorithm. Implementation strategies include dissemination of SPRINT study findings, team-based collaborative care and shared-decision making, blood pressure audit and feedback, home blood pressure monitoring, and health coaching.
  Arms: Intervention

SUMMARY:
The study will test a multifaceted strategy for implementing an intensive blood pressure intervention protocol targeting systolic BP <120 mmHg on cognitive decline in racial minority and low-income hypertensive patients in primary care. The proposed study will generate urgently needed data on effective, adoptable, and equitable intervention strategies to reduce blood pressure-related cognitive decline in low- income and minority populations. If proven effective, the implementation strategy for intensive blood pressure reduction could be adapted and scaled up in diverse primary care settings to prevent cognitive decline and clinical dementia.

DETAILED DESCRIPTION:
African American and low-income populations bear a disproportionate burden of dementia and have been underrepresented in trials of cognitive impairment. The Systolic Blood Pressure Intervention Trial (SPRINT) showed that an intensive blood pressure (BP) intervention (target systolic BP <120 mmHg) lowered the risk of cognitive impairment compared to a standard BP intervention (systolic BP target <140 mmHg). The next important step is to determine how the successful SPRINT intensive blood pressure intervention can be implemented in a real-world clinic setting to prevent cognitive decline. The overall objective of the proposed study is to test a multifaceted strategy for implementing an intensive BP intervention protocol adapted from SPRINT targeting systolic BP <120 mmHg on cognitive decline in racial minority and low-income hypertensive patients in resource-constrained primary care practices in Louisiana and Mississippi. The RE-AIM (Reach Effectiveness Adoption Implementation Maintenance) framework has been used to guide the development and evaluation of the multifaceted implementation strategy, including protocol-based treatment that employs the SPRINT stepped-care intensive BP management algorithm, dissemination of SPRINT findings, shared- decision making, team-based collaborative care, BP audit and feedback, home BP monitoring, and patient health coaching. Building on the ongoing Implementation of Multifaceted Patient-Centered Treatment Strategies for Intensive Blood Pressure Control (IMPACTS-BP) trial, the investigators will cost-effectively conduct a cluster- randomized trial in 40 primary care clinics that serve low-income populations in Louisiana and Mississippi. The primary outcome in the proposed trial is the net difference in mean change of global cognitive composite z-score from baseline to an average of 36 months between the intervention and enhanced usual care groups. Secondary outcomes include net difference in mean change of executive function and memory composite z-scores, systolic and diastolic BP, adverse effects, and quality of life. Implementation outcomes, including acceptability, adaptation, adoption, feasibility, fidelity, penetrance, and cost-effectiveness, will also be collected and used to improve intervention delivery during the trial. The proposed trial, with a sample size of 40 clinics (31.5 patients/clinic), has 93% statistical power to detect a 0.30 or higher difference in the global cognitive composite z-score at a 2-sided significance level of 0.05 assuming 20% loss to follow-up and an intra-cluster correlation of 0.05. In a meta-analysis of 5 clinical trials, the pooled effect size was 0.35 (95% CI 0.32, 0.38) for the global cognitive composite z-score. This study will generate urgently needed data on effective, adoptable, and equitable intervention strategies to reduce blood pressure-related cognitive decline in low-income and minority populations. If proven effective, the implementation strategy for intensive blood pressure reduction could be adapted and scaled up in diverse primary care settings to prevent cognitive decline and clinical dementia.

ELIGIBILITY:
Inclusion Criteria for Primary Care Clinics

* Predominantly managing underserved populations with health disparities (ethnic minorities, low-income groups, and residents of rural areas and inner cities).
* Having electronic medical record systems.
* Serving >200 hypertension patients (ICD-10-CM I10-I15) during the previous year.
* Not participating in other hypertension control programs
* Not sharing providers or nurses/pharmacists with other participating clinics.

Inclusion Criteria for Study Participants

* Men or women aged ≥40 years (2/3 of participants ≥60 years) who receive primary care from participating clinics.
* Systolic BP ≥ 140 mmHg at two screening visits for those not taking antihypertensive medication or systolic BP ≥ 130 mmHg at two screening visits for those taking antihypertensive medications
* Pregnant women, women planning to become pregnant in the near future, women of childbearing potential and not practicing birth control, and persons who cannot give informed consent will be excluded.
* No diagnosis of dementia at baseline
* Baseline MoCA score ≥ 10.
* No diagnosis of end-stage renal disease, defined as dialysis or transplantation
* Speak English as first language
* No plans to change to a primary healthcare provider outside of their clinic in the near future
* No individuals unlikely to complete the study, such as those who plan to move out of the study area in the near future and temporary migrant and homeless people
* No immediate family members are staff at their clinic

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1306 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Net difference in mean change in cognitive decline | Baseline to an average of 36 months
  The net difference in mean change of global cognitive composite z-score over an average 36 months between intervention and enhanced usual care groups

SECONDARY OUTCOMES:
Net difference in mean change in MoCA score | Baseline to an average of 36 months
  Difference between the intervention and usual care group in mean change in Montreal Cognitive Assessment (MoCA) over an average 36 months.
Net difference in mean change in executive function | Baseline to an average of 36 months
  Difference between the intervention and usual care group in mean change in executive function composite z-score (calculated from average of z-scores from individual tests: DSC, Trails A & B, DST, Category Fluency) over an average 36 months.
Net difference in mean change in memory function | Baseline to an average of 36 months
  Difference between the intervention and usual care group in mean change in memory composite z-score (calculated from average of z-scores from individual tests: MoCA immediate & delayed word recall, HVLT-R immediate recall) over an average 36 months.
Net difference in mean change in systolic blood pressure | Baseline to an average of 36 months
  Difference between the intervention and usual care group in mean change in systolic blood pressure over an average 36 months.
Net difference in mean change in diastolic blood pressure | Baseline to an average of 36 months
  Difference between the intervention and usual care group in mean change in diastolic blood pressure over an average 36 months.

OTHER OUTCOMES:
Side effects | Baseline to an average of 36 months
  Difference between the intervention and usual care group in frequency of side effects (collected via detailed questionnaire) over an average 36 months.
Health-related Quality of Life (HRQoL) | Baseline to an average of 36 months
  Difference between the intervention and usual care group in mean change in health-related quality of life (measured using the 12-Item Short Form Survey) over an average 36 months.
Difference in proportion of patients with adjudicated mild cognitive impairment (MCI) or probable dementia (exploratory outcome) | Baseline to an average of 36 months
  Difference in adjudicated MCI and probable dementia at the termination visit between the intervention and usual care group. Based on pre-defined MoCA cutpoints, suspected cases of dementia/MCI will be randomly assigned to two adjudicators, blinded to treatment assignment, with expertise in dementia for review. Data used in the adjudication will include all available cognitive test data, functional assessment, and additional data including demographic information and medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine T Mills, PhD, Principal Investigator — Tulane University; Jiang He, MD, PhD, Principal Investigator — Tulane University; Jeff D Williamson, MD, Principal Investigator — Wake Forest University
Locations (1):
- Tulane University, New Orleans, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Our study data sharing plan will comply with all NIH policies for data sharing. Data sharing will be executed through the centralized NIH data repository and will be implemented in a timely manner. Data will be prepared by the Study Data Coordinating Center and sent to the study's NIA Program Official for review prior to release. These data will be free of identifiers that allow identification of individual research participants either directly or through "deductive disclosure." In addition, the investigators will offer, through our public access website, opportunities for outside investigators to collaborate with us using complete study data.
  At the completion of the project, the investigators will make all intervention materials and procedure manuals available to the public according to the approved plan for making data and materials available to the scientific community, lay public, and the NIH.
Supporting Information: Study Protocol
Time Frame: Study data, including data from baseline and follow-up visits, will be prepared for transmission to the NIH data repository no later than 3 years after the end of the final patient follow-up or 2 years after the main paper of the trial has been published, whichever comes first.